CLINICAL TRIAL: NCT04244006
Title: A Randomized Double-blinded Pilot Study of the Efficacy and Safety of Dupilumab Versus Placebo in Patients With Netherton Syndrome
Brief Title: A Pilot Study of the Efficacy and Safety of Dupilumab Versus Placebo in Patients With Netherton Syndrome
Acronym: NS-DUPI
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Collaborators: MedSharing (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RC31/19/0045
Record Dates: First submitted 2020-01-13; First posted 2020-01-28 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Netherton Syndrome
MeSH Terms: conditions — Netherton Syndrome

STUDY DESIGN:
Intervention Model Description: one arm with dupilumab (2/3 of patients) and one arm with placebo (1/3 of patients)
Who Masked: Participant, Care Provider, Investigator
Masking Description: Dupilumab and placebo will be provided in identically matching 2 mL pre-filled syringes. To protect the blind, each treatment kit of 2 mL (dupilumab/placebo) glass pre-filled syringes will be prepared such that the treatments (dupilumab and its matching placebo) are identical and indistinguishable and will be labeled with a treatment kit number.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dupilumab (Experimental): The patient will receive 2 doses at baseline and then 1 dose every 2 weeks (8 administrations in total) of Dupilumab 300 mg (syringe of 2 mL for subcutaneous administration).
  Interventions: Drug: Dupilumab Prefilled Syringe
- Placebo (Placebo Comparator): The patient will receive 2 doses at baseline and then 1 dose every 2 weeks (8 administrations in total) of placebo (syringe of 2 mL for subcutaneous administration)..
  Interventions: Other: Placebo Prefilled Syringe

INTERVENTIONS:
Drug: Dupilumab Prefilled Syringe — administration of dupilumab corresponding to dupilumab arm
  Arms: Dupilumab
Other: Placebo Prefilled Syringe — administration of placebo corresponding to placebo arm
  Arms: Placebo

SUMMARY:
To date, there are no effective therapy for the management of Netherton Syndrome (NS) Patients use emollients with a limited efficacy on scaling and no efficacy on skin inflammation and pruritus. They may also use topical corticosteroids or calcineurin inhibitors in case of eczematous lesions. The use of therapies targeting skin inflammation has been reported in a few case reports. Their efficacy is very limited and their uses are limited because of the chronicity of the disease, the impaired skin barrier function and the risk for skin infections and skin cancers. Therefore, there is a huge medical need for novel therapies in NS.The expected consequences of this study are that a 16-week course of dupilumab will be more effective than placebo for the treatment of moderate to severe NS Dupilumab could therefore improve skin condition and quality of life.

DETAILED DESCRIPTION:
This is a proof of concept (pilot) double-blind randomized placebo-controlled study evaluating the efficacy and safety of dupilumab for the treatment of NS. Patients will be randomized in a 2:1 ratio to receive dupilumab (2 doses of 300 mg), or placebo, at baseline and then 1 dose of dupilumab 300 mg, or placebo, every 2 weeks until week 14 (total of 8 administrations).Moderate to severe NS were selected in order to be able to measure the improvement of skin condition.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients affiliated to a social insurance protection regimen.
* Clinical diagnosis of NS (7) (trichorrhexis invaginata, extensive scaling, skin inflammation, allergic manifestations) and absent or marked reduction of LEKTI staining.
* Moderate to severe forms: NASA (Netherton Area Severity Assessment score) score ≥ 5/12 at inclusion.
* Patients able to understand the study procedures including the ability to complete patient-based self-assessment questionnaires.
* Patients who agree to sign the written informed consent.

Exclusion Criteria:

* Hypersensitivity to dupilumab or its excipients.
* Modification of the usual treatment (emollients and topical corticosteroids used on a regular basis) within 2 weeks before inclusion.
* Treatment with topical calcineurin inhibitors 1 week before inclusion.
* Treatment with oral immunosuppressant (including cyclosporine, methotrexate, azathioprine, mycophenolate mofetil), oral retinoids (acitretin, alitretinoin, isotretinoin) or phototherapy within 4 weeks before inclusion.
* Treatment with immunomodulating biologics (Tumor Necrosis Factor (TNF) inhibitor) 16 weeks before inclusion.
* Treatment with another investigational drug within 8 weeks before inclusion.
* Treatment with a systemic antibiotic within 2 weeks before inclusion.
* Active skin infection requiring the use of a systemic therapy within 2 weeks before the inclusion.
* Any other condition that according to the investigator will impair the ability to evaluate treatment effect.
* Known or suspected history of immunosuppression, including history of invasive opportunistic infections (e.g., tuberculosis, histoplasmosis, listeriosis, coccidioidomycosis, pneumocystis, aspergillosis).
* Current infections including infection with helminthes.
* Pregnant or breastfeeding women, or women planning to become pregnant or breastfeed during the study. Women of childbearing age, potentially sexually active, and unwilling to use adequate birth control methods.
* Mental or physical incapacity to fill in the questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-07-23 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
The severity of the disease of the Netherton Area Severity Assessment score (NASA). | Day 0 and week 16
  NASA score

SECONDARY OUTCOMES:
Clinical efficacy severity of pruritus and pain | Day 0, week 2, week 4, week 6, week 8, week 10, week 12, week 14, week 16, week 28
  NASA score
Presence of infections (adverse event) | Day 0, week 2, week 4, week 6, week 8, week 10, week 12, week 14, week 16, week 28
  Number of Bacterial or viral Skin infections
Quantity of dermocorticosteroids used between each visit will be evaluated by questioning the patient. | Day 0, week 2, week 4, week 6, week 8, week 10, week 12, week 14, week 16, week 28
  number of tubes multiplied by the weight of one tube
QOL score | Day 0, Week 16 and 28
  QOL score
Skin inflammation | Day 0 and week 16
  number of inflammation markers on biopsies
Protease activity | Day 0 and week 16
  number of protease markers on biopsies
Microbiome qualitative and quantitative analysis | Day 0 and week 16
  number and form of bacteria
Transepidermal water loss (TEWL) | Day 0 and Week 16
  Measured by a Tewameter applied on a standardized area in the anterior aspect of the forearm,
Safety of dupilumab | Day 0, week 2, week 4, week 6, week 8, week 10, week 12, week 14, week 16, week 28
  Blood tests performed every month until Week 16 (liver and renal tests, total blood count)

CONTACTS AND LOCATIONS:
Overall Officials: Juliette MAZEREEUW-HAUTIER, Principal Investigator — Toulouse Hospital
Locations (2):
- France (2):
  - Dermatologie Necker, Paris
  - Dermatology, Toulouse

IPD SHARING:
Plan to Share IPD: No